CLINICAL TRIAL: NCT05298566
Title: Factors Affecting Quality of Life in Patient With Chronic Musculoskeletal Pain
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Tugba Sahbaz, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: KAEK/2021.11.306
Record Dates: First submitted 2022-02-03; First posted 2022-03-28 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Quality of Life; Chronic Musculoskeletal Disease; Chronic Pain
Keywords: quality of life; disabilty; Chronic musculoskeletal pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study included patients who applied to the physical therapy and rehabilitation outpatient clinic and were diagnosed with chronic low back pain and osteoarthrosis and met the criteria for participation in the study.

Demografik datas, pain , Functional Limitations and Quality of Life wa evaluated.

DETAILED DESCRIPTION:
When treating diseases, clinicians traditionally aim for pain reduction and functional recovery. This is also true for chronic musculoskeletal diseases. However, the psychosocial support required to improve the general health perception of patients is becoming increasingly important. In clinical practice, it is essential to evaluate the quality of life and general well-being and to evaluate the patient completely biopsychosocially . Determining the factors affecting the quality of life is important in terms of contributing to the rehabilitation processes and treatment plans of CMP patients. In this direction, our study aims to examine the factors affecting the quality of life.

When treating diseases, clinicians traditionally aim for pain reduction and functional recovery. This is also true for chronic musculoskeletal diseases. However, the psychosocial support required to improve the general health perception of patients is becoming increasingly important. In clinical practice, it is essential to evaluate the quality of life and general well-being and to evaluate the patient completely biopsychosocially . Determining the factors affecting the quality of life is important in terms of contributing to the rehabilitation processes and treatment plans of CMP patients. In this direction, our study aims to examine the factors affecting the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years old
* Clinical diagnosis of spondilosis and gonarthrosis-
* Must not be surgical indication

Exclusion Criteria:

* History of knee or back surgery
* Detection of muscle weakness on physical examination
* Presence of additional neurological disease that will affect the patient's mobilization and cognitive level
* Presence of Cognitive impairment
* Presence of Chronic pain of nonmusculoskeletal origin (gynocological, retroperitoneal, abdominal)
* Being treated for depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients who applied to the physical therapy and rehabilitation outpatient clinic and were diagnosed with chronic low back pain and osteoarthrosis and meeting the criteria for participation in the study will be included in our study.
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2022-03-27 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Pain Severity | Baseline
  The severity of rest pain and activity pain experienced by the patients in the last 1 week will be evaluated by VAS, which is a numeric rating scale. The highest pain intensity is 10, o no pain, 5 will be scored as moderate pain. Higher scores mean more pain intensity
Functioal Limitation | baseline
  Roland Morris questionare (RMQ) will be used for disability assessment in patients with chronic low back pain.Roland Morris questionare evaluates functional limitation due to low back pain. The total maximum score is 24. It includes a total of 24 items questioning patients' mobility, self-care and sleep status.
  Disability in patients with knee osteoarthritis will be evaluated with the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC).WOMAC; It is a 24-item scale that examines three dimensions: pain, stiffness and physical function. Higher scores mean more disability
Health-related quality of life | Baseline
  The Short Form Health Questionnaire (SF-36) questionnaire, which examines health-related quality of life under eight sub-titles; It consists of 36 items. The SF36 questionnaire will be used in the study.

CONTACTS AND LOCATIONS:
Overall Officials: Tugba Sahbaz, MD, Study Director — Kanuni Sultan Suleyman Research Hospital
Locations (1):
- kanuni Sultan suleyman Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeong H, Lee Y. Sex-Based Differences in the Quality of Life of Elderly Koreans with Chronic Musculoskeletal Pain. Int J Environ Res Public Health. 2020 Jan 23;17(3):743. doi: 10.3390/ijerph17030743. PMID 31979306
- [Background] Agnus Tom A, Rajkumar E, John R, Joshua George A. Determinants of quality of life in individuals with chronic low back pain: a systematic review. Health Psychol Behav Med. 2022 Jan 5;10(1):124-144. doi: 10.1080/21642850.2021.2022487. eCollection 2022. PMID 35003902
- [Background] Koçyiğit H AÖ FG. Kısa Form-36'nın Türkçe versiyonunun güvenlirliği ve geçerliliği. İlaç ve Tedavi Dergisi (12):102-6.
- [Background] Basaran S, Guzel R, Seydaoglu G, Guler-Uysal F. Validity, reliability, and comparison of the WOMAC osteoarthritis index and Lequesne algofunctional index in Turkish patients with hip or knee osteoarthritis. Clin Rheumatol. 2010 Jul;29(7):749-56. doi: 10.1007/s10067-010-1398-2. Epub 2010 Feb 19. PMID 20169459